







## **INFORMED CONSENT FORM**

**Tuberculosis screening with AeoNose and CAD4TB in Paraguayan prisons** 

**PriNose Study** 

December 2019

## **INFORMED CONSENT**

I was invited to participate in the study to diagnose tuberculosis.

I understand that I must perform a standardized routine that was previously shown to me by video and I must allow researchers to monitor my clinical, radiological, and laboratory status and I will breathe through an electronic nose device for 5 minutes.

I authorize the exchange of all test results between the research team and the National Tuberculosis Control Program (PNCT). I am aware that in the event of a positive result for tuberculosis an immediate initiation of treatment supervised by the PNCT will be offered.

I have been informed of the benefits for myself and my family members and that I will not receive financial rewards. I have been provided with the name of an independent target staff who can be easily contacted to answer my questions.

I read the consent form provided or it was read to me. I had the opportunity to ask about it and the questions have been answered satisfactorily.

I give my voluntary consent to participate in this research and understand that I have the right to withdraw from the research at any time without, in any way, affecting my medical care.

| Name of subject: | |
|---|---|
| Signature / fingerprint: | Fingerprint |
| I certify that I have fully informed this subject about the study. | |
| Name of investigator (or his/her representative): | |
| Signature: Date: / / | |
| Additional information was provided by (witness): | |
| Name: | |
| Function: | |
| Signature: | |

The subject will receive a signed version of the informed consent form.